CLINICAL TRIAL: NCT02514239
Title: An Open Label, Phase I, Dose Escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Doses of BI 836909 in Relapsed and/or Refractory Multiple Myeloma Patients
Brief Title: Phase I Dose Escalation of i.v. BI 836909 Monotherapy in Last Line Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1351.1; 2014-004896-22 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-08-03 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

ARMS (13):
- Intravenous Infusion of BI 836909 (0.2 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (0.4 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (0.8 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (1.6 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (3.2 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (6.5 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (13 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (25 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (50 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (100 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (200 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (400 μg/d) (Experimental)
  Interventions: Drug: BI 836909
- Intravenous Infusion of BI 836909 (800 μg/d) (Experimental)
  Interventions: Drug: BI 836909

INTERVENTIONS:
Drug: BI 836909 — Intravenous Infusion of BI 836909.
  Other Names: AMG 420

SUMMARY:
The primary objective of this trial is to determine the maximum tolerated dose (MTD) of BI 836909 administered by continuous i.v. infusion in patients with relapsed and/or refractory multiple myeloma. If the MTD is not reached based on safety findings, a recommended dose for further development will be determined. This will depend on the safety data, pharmacokinetic/pharmacodynamics data and potentially preliminary efficacy data. Secondary objectives are to document the safety and tolerability of BI 836909, to perform pharmacokinetic and pharmacodynamic analyses and to evaluate relevant biological effects in terms of parameters of efficacy.

ELIGIBILITY:
Inclusion criteria:

* Patients with a documented diagnosis of relapsed and/or refractory multiple myeloma who progressed after at least two prior treatment regimens, including both proteasome inhibitor as well as an immune-modulatory drug at time of screening
* must have measurable disease, defined by one or more of following at time of screening:

  * a serum M protein > 0.5 g/dl measured by serum protein electrophoresis
  * urinary M protein excretion > 200 mg/24 hours
  * serum free light chain (FLC) measurement > 10 mg/dl, provided that the serum FLC ratio is abnormal
* Relapse or progression of disease with an indication for therapy as per investigator´s judgement at time of screening
* ECOG Performance Status 0, 1 or 2 at time of screening
* Age >= 18 years at time of screening
* Written informed consent which is consistent with ICH_GCP guidelines and local legislation
* Able to adhere to the study visit schedule e.g. ability to come to the clinic and to other protocol requirements
* Indwelling central venous catheter or willingness to undergo intra venous central line placement.

Exclusion criteria:

* Plasma cell leukemia
* Extramedullary relapse of multiple myeloma
* Known central nervous system involvement by multiple myeloma
* Last anticancer treatment < 2 weeks prior to visit 1
* Last treatment with a therapeutic antibody less than 6 weeks prior to visit 1
* Prior allogeneic stem cell transplantation or solid organ transplantation
* Autologous bone marrow transplantation < than 90 days at time of treatment start
* Last corticosteroid < 2 weeks prior to visit 1 unless the dose is <= 10 mg/day prednisolone or equivalent
* AST or ALT > 3 x upper limit of normal (CTCAE version 4.03 grade 2 or higher) at time of screening
* Total conjugated bilirubin > 1.5 x upper limit of normal (CTCAE version 4.03 grade 2 or higher) at time of screening
* Absolute neutrophil count < 1.0 x 109/L (without growth factor support) at time of screening
* Platelets < 25 x 109/L (without transfusions) at time of screening
* Calculated GFR < 30 mL/min (Cockcroft-Gault Formula) at time of screening
* Clinical relevant concurrent medical disease or condition which according to the investigator's judgement would either compromise patient safety or interfere with the evaluation of the safety of the test drug, e.g. symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy at time of screening
* clinically not controlled chronic or ongoing infectious disease requiring treatment at the time of enrolment or within the previous two weeks
* Active hepatitis B or C, or laboratory evidence for a chronic infection with hepatitis B or C at time of screening; HIV infection at time of screening
* Women of childbearing potential not using highly effective method of birth control during the trial until one year after the last dose. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year)when used consistently and correctly used such as implants, injectables, combined oral contraceptives, intrauterine devises (IUDs), sexual abstinence or vasectomised partner. Barrier methods of contraception are accepted if condom or occlusive cap is used together with spermicides (e.g. foam, gel). Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation/salpingectomy, or postmenopausal (12 months with no menses without an alternative medical cause
* Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second medically acceptable method of contraception during the trial and for a minimum of 6 months after treatment
* Pregnancy or breast feeding
* Known or suspected active alcohol or drug abuse as per investigator's judgement
* Treatment with another investigational drug within the past four weeks before start of therapy or concomitantly with this trial
* Patients with known hypersensitivity to any component of the study drug
* Patients with other malignancies within 5 years at time of screening (except basal cell or squamous cell carcinoma of the skin or carcinoma in situ treated with curative therapy)
* Known autoimmune diseases requiring systemic treatment in past 5 years and interfering with evaluation of study drug
* Pre-existing disorders of the central nervous system

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- France (3):
  - HOP Claude Huriez, Lille
  - HOP Hôtel-Dieu, Nantes
  - INS Universitaire du Cancer, Toulouse
- Germany (2):
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Topp MS, Duell J, Zugmaier G, Attal M, Moreau P, Langer C, Kronke J, Facon T, Salnikov AV, Lesley R, Beutner K, Kalabus J, Rasmussen E, Riemann K, Minella AC, Munzert G, Einsele H. Anti-B-Cell Maturation Antigen BiTE Molecule AMG 420 Induces Responses in Multiple Myeloma. J Clin Oncol. 2020 Mar 10;38(8):775-783. doi: 10.1200/JCO.19.02657. Epub 2020 Jan 2. PMID 31895611
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, non-randomised, phase I, dose escalation trial in patients with relapsed and/or refractory multiple myeloma. The first 4 dose levels (0.2, 0.4,0.8, and 1.6 Microgram Per Day (μg/d)) were tested in single patient cohorts. Dose levels ≥3.2 μg/d (3.2, 6.5, 13, 25, 50, 100, 200, 400, and 800 μg/d) were to be tested in a 3+3 design. Once the Maximum tolerated dose (MTD) was determined, up to 6 additional patients were to be treated at the MTD or at the recommended dose.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d): Intravenous infusion of BI 836909 (overall in the 4 lowest dose cohorts 0.2, 0.4, 0.8, 1.6 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (3.2 μg/d): Intravenous infusion of BI 836909 (3.2 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (6.5 μg/d): Intravenous infusion of BI 836909 (6.5 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (13 μg/d): Intravenous infusion of BI 836909 (13 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (25 μg/d): Intravenous infusion of BI 836909 (25 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (50 μg/d): Intravenous infusion of BI 836909 (50 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (100 μg/d): Intravenous infusion of BI 836909 (100 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (200 μg/d): Intravenous infusion of BI 836909 (200 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (400 μg/d): Intravenous infusion of BI 836909 (400 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (800 μg/d): Intravenous infusion of BI 836909 (800 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
Period: Overall Study
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Started | 5 | 4 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Treated | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Completed (10 cycles completed) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not Completed | 5 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 8 | 3
Not completed — Refused to continue trial medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Dose-limiting toxicity (DLT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Adverse Events | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Not completed — Progressive disease | 3 | 3 | 2 | 2 | 3 | 3 | 4 | 2 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients who were administered trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d) | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.3) | 67.7 (2.5) | 63.0 (9.8) | 69.3 (6.1) | 67.0 (7.5) | 61.6 (4.6) | 62.5 (7.8) | 62.7 (14.5) | 57.7 (12.2) | 71.3 (8.6) | 62.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 1 | 3 | 3 | 15
  Male | 4 | 1 | 3 | 2 | 2 | 2 | 4 | 2 | 7 | 0 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 1 | 3 | 2 | 2 | 3 | 2 | 2 | 8 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of BI 836909
Description: The Maximum tolerated dose (MTD) of BI 836909, which was defined as the highest dose of the dose level tested where ≤1 patient out of 6 developed a Dose-limiting toxicity (DLT). The MTD was defined based on DLTs observed during Cycle 1. However, all Adverse Events corresponding to the definition of a DLT (see below) were to be considered for confirming the MTD. A DLT was defined as any drug-related non-haematological Adverse Event of Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade 3 or higher.
Time Frame: Cycle 1, up to 6 weeks.
Population: MTD evaluation set (MTDS): all patients who were administered trial medication and who were not replaced for the Maximum tolerated dose (MTD) determination.
Measure: Number; unit: Microgram Per Day (μg/d)
Groups:
- Intravenous Infusion of BI 836909 (Total Dose Escalation): BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable Adverse Events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles. The first 4 dose levels (0.2, 0.4,0.8, and 1.6 Microgram Per Day (μg/d)) were tested in single patient cohorts. Dose levels ≥3.2 μg/d (3.2, 6.5, 13, 25, 50, 100, 200, 400, and 800 μg/d) were tested in a 3+3 design.
Arm/Group | Intravenous Infusion of BI 836909 (Total Dose Escalation)
Number analyzed (Participants) | 34
Microgram Per Day (μg/d) | 400

2. Primary Outcome: The Number of Patients With Dose-limiting Toxicities (DLTs)
Description: The number of patients with Dose-limiting toxicities (DLTs) in cycle 1. A Dose-limiting toxicity was defined as any drug-related non-haematological Adverse Event of Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade 3 or higher.
Time Frame: Cycle 1, up to 6 weeks.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

3. Secondary Outcome: Number of Participants With an Objective Response
Description: Objective responses: Stringent complete response (sCR): CR + normal Free light chain (FLC) ratio and no clonal cells in bone marrow by immunohistochemistry or immunofluorescence. CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow. Very good partial response (VGPR): serum and urine M protein detectable by immunofixation but not on electrophoresis or >90% reduction in serum M protein plus urine M protein level <100 mg/24h. PR: >50% reduction of serum and 24 h urinary M protein by >90% or to <200mg/24h. If unmeasurable, a >50% decrease in difference between involved and uninvolved FLC levels instead of M protein criteria. if FLC assay was not measurable, a >50% reduction in plasma cells was required instead of M protein, provided baseline bone marrow plasma cell was >30%. In addition to the listed criteria, a >50% reduction in the size of soft tissue plasmacytomas was also required, if present at baseline.
Time Frame: On-treatment: From start of treatment till end of trial (EOT) visit, up to 61 weeks. Extended follow-up: From start of treatment till the last extended follow-up visit which was scheduled at 12 months after end of treatment, up to 113 weeks.
Population: Treated set (TS): all patients who were administered trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Participants
  On treatment: Stringent complete response (sCR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0
  On treatment: Complete response (CR) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  On treatment: Very good partial response (VGPR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  On treatment: Partial response (PR) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  On treatment: No response (stable disease or disease progression) | 5 | 3 | 2 | 3 | 3 | 4 | 3 | 2 | 3 | 1
  On treatment + extended follow-up visits (follow-up: Stringent complete response (sCR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0
  On treatment + extended follow-up visits (follow-up: Complete response (CR) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  On treatment + extended follow-up visits (follow-up: Very good partial response (VGPR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  On treatment + extended follow-up visits (follow-up: Partial response (PR) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  On treatment + extended follow-up visits (follow-up: No response (stable disease or disease progression) | 5 | 3 | 2 | 3 | 3 | 4 | 3 | 2 | 3 | 1

4. Secondary Outcome: Duration of Objective Response - on Treatment
Description: For patients with objective response, the duration of response was calculated from the time of first recorded achievement of a response (sCR, CR, PR, or VGPR) until documented progression or death. The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From start of treatment till end of trial (EOT) visit, up to 61 weeks.
Population: All patients who were administered trial medication and showed an objective response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 7 | 2
Months |  |  | NA [NA to NA] — Insufficient number of participants with events. |  |  | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [4.63 to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Insufficient number of participants with events.

5. Secondary Outcome: Duration of Objective Response - Including Extended Follow up Visits
Description: as for outcome 4
Time Frame: From start of treatment till the last extended follow-up visit which is scheduled at 12 months after end of treatment, up to 113 weeks.
Population: All patients who were administered trial medication and showed an objective response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 7 | 2
Months |  |  | NA [NA to NA] — Insufficient number of participants with events. |  |  | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | 23.62 [4.63 to 24.18] | NA [NA to NA] — Insufficient number of participants with events.

6. Secondary Outcome: Number of Participants With a Minimal Residual Disease (MRD) Response
Description: Minimal residual disease (MRD) response was defined as <1 tumour cell within 10000 normal cells in bone marrow. MRD was determined using Fluorescence-activated cell sorting (FACS) analysis.
Time Frame: On-treatment: From start of treatment till end of trial (EOT) visit, up to 61 weeks. Follow-up: From start of treatment till the last extended follow-up visit which was scheduled at 12 months after end of treatment, up to 113 weeks.
Population: Treated set (TS): all patients who were administered trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Participants
  On treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 0
  On treatment + extended follow-up visits (follow-up) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 0

7. Secondary Outcome: Duration of Minimal Residual Disease (MRD) Response - on Treatment
Description: Duration of MRD response was calculated from the time of first recorded achievement of a MRD response to documented progression or death. The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From start of treatment till end of trial (EOT) visit, up to 61 weeks.
Population: All patients who were administered trial medication and showed a Minimal residual disease (MRD) response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 0
Months |  |  | NA [NA to NA] — Insufficient number of participants with events. |  |  |  |  | NA [NA to NA] — Insufficient number of participants with events. | NA [9.00 to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. |

8. Secondary Outcome: Duration of Minimal Residual Disease (MRD) Response - Including Extended Follow up Visits
Description: as for outcome 7
Time Frame: From start of treatment till the last extended follow-up visit which was scheduled at 12 months after end of treatment, up to 113 weeks.
Population: All patients who were administered trial medication and showed a Minimal residual disease (MRD) response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 0
Months |  |  | NA [NA to NA] — Insufficient number of participants with events. |  |  |  |  | NA [NA to NA] — Insufficient number of participants with events. | 20.70 [9.00 to 22.77] |

9. Secondary Outcome: Progression-free Survival (PFS) - on Treatment
Description: PFS was defined as time from first treatment with BI 836909 till disease progression or death. Progression was defined according to International Myeloma Working Group (IMWG 2006) response criteria as an increase >25% from lowest response value in any of the following parameters: -Serum M protein (absolute increase had to be >0.5 gram/ deciliters (dL)) -Urine M protein (absolute increase had to be >200 milligram (mg)/24 hour) -Only in patients without measurable serum and urine M protein levels The difference between involved and uninvolved FLC levels. Absolute increase had to be >10 mg/dL -Bone marrow plasma cell percentage; absolute percentage had to be >10% -Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas -Development of hypercalcaemia (corrected serum calcium >11.5 mg/dL or 2.65 Millimole/Liter) that was attributed solely to the plasma cell proliferative disorder.
Time Frame: From start of treatment till end of trial (EOT) visit, up to 61 weeks.
Population: Treated set (TS): all patients who were administered trial medication.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Months | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | 5.55 [0.95 to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial.

10. Secondary Outcome: Progression-free Survival (PFS) - Including Extended Follow up Visits
Description: as for outcome 9
Time Frame: as for outcome 8
Population: Treated set (TS): all patients who were administered trial medication.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Intravenous Infusion of BI 836909 (Overall in the 4 Lowest Dose Cohorts 0.2, 0.4, 0.8, 1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 10 | 3
Months | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial. | 7.74 [0.95 to 24.41] | NA [NA to NA] — Estimates for median and/or IQR are missing because the largest observation was censored and the estimation was restricted to the largest event time observed in this clinical trial.

11. Secondary Outcome: Serum Concentration at Steady State of BI 836909 (Css)
Description: Serum concentration at steady state of BI 836909 (Css).
Time Frame: Pharmacokinetic samples were collected at 48:00 hours (h):minutes (min), 168:00, 336:00, 504:00 and 671:50 h after the start of infusion of BI 836909 of the first cycle.
Population: PK Analysis Set (PKS): all evaluable patients in the treated set which provide at least one evaluable observation for at least one PK endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Groups:
- Intravenous Infusion of BI 836909 (0.2 μg/d): Intravenous infusion of BI 836909 (0.2 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (0.4 μg/d): Intravenous infusion of BI 836909 (0.4 Microgram Per Day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable Adverse Events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (0.8 μg/d): Intravenous infusion of BI 836909 (0.8 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
- Intravenous Infusion of BI 836909 (1.6 μg/d): Intravenous infusion of BI 836909 (1.6 microgram per day (μg/d)). BI 836909 was administered as 4-week continuous intravenous infusion (c.i.v.) followed by a 2-week treatment break for 5 cycles or until progression, unacceptable adverse events, or any other reason necessitating withdrawal. In case of ongoing clinical benefit and if considered indicated by the investigator, 5 additional treatment cycles could be done, leading to a maximum of 10 cycles.
Arm/Group | Intravenous Infusion of BI 836909 (0.2 μg/d) | Intravenous Infusion of BI 836909 (0.4 μg/d) | Intravenous Infusion of BI 836909 (0.8 μg/d) | Intravenous Infusion of BI 836909 (1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 9 | 2
picogram/milliliter (pg/mL) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the serum concentrations of BI 836909 were below limit of quantitation (BLQ) for 0.2 ug/day. | 86.5 (NA) — Geometric Coefficient of Variation could not be calculated because of the limited sample size. | 90.8 (41.1) | 184 (NA) — Geometric Coefficient of Variation could not be calculated because of the limited sample size. | 526 (34.7) | 1070 (67.3) | 2180 (34.6) | 4130 (30.7) | 10700 (55.4) | 9810 (47.6) | 14100 (121) | 29900 (54.3) | 33000 (41.0)

ADVERSE EVENTS:
Time Frame: Adverse Events collected from start of treatment till the last day of treatment + 30 Residual Effect Period, up to 436 days. All-cause Mortality collected from start of treatment till the last follow up visit, up to 113 weeks.
Description: Treated set (TS): all patients who were administered trial medication.
Arm/Group | Intravenous Infusion of BI 836909 (0.2 μg/d) | Intravenous Infusion of BI 836909 (0.4 μg/d) | Intravenous Infusion of BI 836909 (0.8 μg/d) | Intravenous Infusion of BI 836909 (1.6 μg/d) | Intravenous Infusion of BI 836909 (3.2 μg/d) | Intravenous Infusion of BI 836909 (6.5 μg/d) | Intravenous Infusion of BI 836909 (13 μg/d) | Intravenous Infusion of BI 836909 (25 μg/d) | Intravenous Infusion of BI 836909 (50 μg/d) | Intravenous Infusion of BI 836909 (100 μg/d) | Intravenous Infusion of BI 836909 (200 μg/d) | Intravenous Infusion of BI 836909 (400 μg/d) | Intravenous Infusion of BI 836909 (800 μg/d) | Intravenous Infusion of BI 836909 (Total Dose Escalation)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/1 | 0/3 | 0/3 | 0/3 | 0/3 | 1/5 | 0/4 | 0/3 | 1/10 | 0/3 | 2/42
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/2 | 0/1 | 1/3 | 3/3 | 1/3 | 1/3 | 3/5 | 2/4 | 3/3 | 8/10 | 3/3 | 27/42
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/2 | 1/1 | 3/3 | 3/3 | 3/3 | 3/3 | 5/5 | 4/4 | 3/3 | 10/10 | 2/3 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Infusion of BI 836909 (0.2 μg/d) (N=1) | Intravenous Infusion of BI 836909 (0.4 μg/d) (N=1) | Intravenous Infusion of BI 836909 (0.8 μg/d) (N=2) | Intravenous Infusion of BI 836909 (1.6 μg/d) (N=1) | Intravenous Infusion of BI 836909 (3.2 μg/d) (N=3) | Intravenous Infusion of BI 836909 (6.5 μg/d) (N=3) | Intravenous Infusion of BI 836909 (13 μg/d) (N=3) | Intravenous Infusion of BI 836909 (25 μg/d) (N=3) | Intravenous Infusion of BI 836909 (50 μg/d) (N=5) | Intravenous Infusion of BI 836909 (100 μg/d) (N=4) | Intravenous Infusion of BI 836909 (200 μg/d) (N=3) | Intravenous Infusion of BI 836909 (400 μg/d) (N=10) | Intravenous Infusion of BI 836909 (800 μg/d) (N=3) | Intravenous Infusion of BI 836909 (Total Dose Escalation) (N=42)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 5
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Infusion of BI 836909 (0.2 μg/d) (N=1) | Intravenous Infusion of BI 836909 (0.4 μg/d) (N=1) | Intravenous Infusion of BI 836909 (0.8 μg/d) (N=2) | Intravenous Infusion of BI 836909 (1.6 μg/d) (N=1) | Intravenous Infusion of BI 836909 (3.2 μg/d) (N=3) | Intravenous Infusion of BI 836909 (6.5 μg/d) (N=3) | Intravenous Infusion of BI 836909 (13 μg/d) (N=3) | Intravenous Infusion of BI 836909 (25 μg/d) (N=3) | Intravenous Infusion of BI 836909 (50 μg/d) (N=5) | Intravenous Infusion of BI 836909 (100 μg/d) (N=4) | Intravenous Infusion of BI 836909 (200 μg/d) (N=3) | Intravenous Infusion of BI 836909 (400 μg/d) (N=10) | Intravenous Infusion of BI 836909 (800 μg/d) (N=3) | Intravenous Infusion of BI 836909 (Total Dose Escalation) (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 2 | 1 | 5 | 1 | 15
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 5
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth demineralisation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 5
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 6
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 11
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 7 | 2 | 12
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 6
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4
Eosinophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 2 | 2 | 5 | 2 | 23
Monocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 5 | 1 | 10
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 2 | 10
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 6 | 2 | 16
pH urine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 5 | 2 | 13
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tongue paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02514239/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02514239/SAP_001.pdf